CLINICAL TRIAL: NCT06109714
Title: Early Biomarker Kidney Injury Assessment After Acumen Directed Fluid Management in Cardiac Surgery
Acronym: BE-KIND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Reney Henderson, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HP-00100950
Record Dates: First submitted 2022-06-01; First posted 2023-10-31 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Renal Injury; Acute Kidney Injury
Keywords: Cardiac Surgery; Cardiac Surgery Induced Kidney Injury; Kidney Biomarkers
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACUMEN guided resuscitation protocol (Experimental): Fluid resuscitation and hemodynamic management will be guided by ACUMEN based off a protocol.
  Interventions: Other: Goal Directed Fluid Therapy
- Standard of care resuscitation (No Intervention): Fluid resuscitation will be guided by standard monitors (urine output, blood loss, transesophageal echocardiography).

INTERVENTIONS:
Other: Goal Directed Fluid Therapy — Fluid administration and hemodynamic management guided with the assistance of Edwards Lifesciences ACUMEN monitor
  Arms: ACUMEN guided resuscitation protocol

SUMMARY:
This study is to assess the benefits of goal-directed fluid management with ACUMEN in cardiac surgical patients and its impact on cardiac surgery-induced kidney injury.

DETAILED DESCRIPTION:
This study is to assess the benefits of goal-directed fluid management with ACUMEN in cardiac surgical patients undergoing a CABG, AVR, or CABG/AVR. Kidney injury biomarkers NGAL, Uromodulin, and Hepcidin-25 will be used to assess cardiac-induced kidney injury. Patients will be randomly enrolled in either standard care for fluid management or goal-directed fluid management with ACUMEN.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing cardiopulmonary bypass
* Procedure coronary artery bypass grafting, aortic valve replacement, or both

Exclusion Criteria:

* Patients < 18 years old
* Emergent surgery
* Preoperative kidney disease (Cr > 2.0 or on renal replacement therapy)
* Ejection fraction < 40%
* Incomplete data in medical record

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury | 7 days or discharge whichever occurs first
  KIDIGO Criteria for AKI
Renal Biomarkers | 48 hours postoperatively
  NGAL, Hepcidin-25, and Uromodulin

SECONDARY OUTCOMES:
Total Fluid Administered | From initiation of surgery to 48 hours postoperatively
  intraoperative and postoperative volume given measured in milliliters
ICU Length of Stay | From admission to the intensive care unit until discharge or 20 weeks whichever comes first.
  Quantified in days and hours
Hemodynamic Support Usage | During the first 48 hours postoperatively
  Vasopressor or Inotrope usage
Morbidity and Mortality | 30 days
  Death and Major adverse events (cerebral vascular stroke, myocardial infarction, infection, prolonged intubation > 24 hours)
Blood Transfusions | From surgical incision to 48 hours postoperatively
  Any Allogeneic Blood Transfusions

CONTACTS AND LOCATIONS:
Overall Officials: Reney A Henderson, MD, Principal Investigator — University of Maryland, Baltimore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kullmar M, Massoth C, Ostermann M, Campos S, Grau Novellas N, Thomson G, Haffner M, Arndt C, Wulf H, Irqsusi M, Monaco F, Di Prima A, Garcia Alvarez M, Italiano S, Cegarra SanMartin V, Kunst G, Nair S, L'Acqua C, Hoste EAJ, Vandenberghe W, Honore PM, Kellum J, Forni L, Grieshaber P, Weiss R, Gerss J, Wempe C, Meersch M, Zarbock A. Biomarker-guided implementation of the KDIGO guidelines to reduce the occurrence of acute kidney injury in patients after cardiac surgery (PrevAKI-multicentre): protocol for a multicentre, observational study followed by randomised controlled feasibility trial. BMJ Open. 2020 Apr 6;10(4):e034201. doi: 10.1136/bmjopen-2019-034201. PMID 32265240
- [Background] Vives M, Hernandez A, Parramon F, Estanyol N, Pardina B, Munoz A, Alvarez P, Hernandez C. Acute kidney injury after cardiac surgery: prevalence, impact and management challenges. Int J Nephrol Renovasc Dis. 2019 Jul 2;12:153-166. doi: 10.2147/IJNRD.S167477. eCollection 2019. PMID 31303781
- [Background] Van den Eynde J, Schuermans A, Verbakel JY, Gewillig M, Kutty S, Allegaert K, Mekahli D. Biomarkers of acute kidney injury after pediatric cardiac surgery: a meta-analysis of diagnostic test accuracy. Eur J Pediatr. 2022 May;181(5):1909-1921. doi: 10.1007/s00431-022-04380-4. Epub 2022 Jan 17. PMID 35039910
- [Background] Nadim MK, Forni LG, Bihorac A, Hobson C, Koyner JL, Shaw A, Arnaoutakis GJ, Ding X, Engelman DT, Gasparovic H, Gasparovic V, Herzog CA, Kashani K, Katz N, Liu KD, Mehta RL, Ostermann M, Pannu N, Pickkers P, Price S, Ricci Z, Rich JB, Sajja LR, Weaver FA, Zarbock A, Ronco C, Kellum JA. Cardiac and Vascular Surgery-Associated Acute Kidney Injury: The 20th International Consensus Conference of the ADQI (Acute Disease Quality Initiative) Group. J Am Heart Assoc. 2018 Jun 1;7(11):e008834. doi: 10.1161/JAHA.118.008834. No abstract available. PMID 29858368